CLINICAL TRIAL: NCT04552691
Title: Expanded Access Treatment With Open-Label Pegunigalsidase Alfa for Fabry Patients
Brief Title: Open-Label Expanded Access Treatment With Pegunigalsidase Alfa for Fabry Disease Patients
Status: Approved for marketing | Type: Expanded Access
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Chiesi USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-102-F90
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; Pegunigalsidase alfa
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Pegunigalsidase Alfa — Pegunigalsidase alfa is a recombinant ERT (enzyme replacement therapy) used to treat Fabry disease (dosage: 1 mg/kg body weight every 2 weeks).

SUMMARY:
The objective of this treatment protocol is to provide guidance to Treating Physicians who seek access to pegunigalsidase alfa for Fabry patients whose clinical condition, in the opinion of the Treating Physician, requires treatment with enzyme replacement therapy (ERT) with pegunigalsidase alfa and a) cannot be adequately treated with currently approved FDA products and/or b) are not able or willing to participate in any of the on-going clinical trials in the United States.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the Treating Physician, the patient cannot be adequately treated with any FDA approved drugs for Fabry and is not able to enroll in any current clinical trial for Fabry disease.
* Patient (or legal guardian) is able to sign an informed consent prior to treatment.
* A documented diagnosis of Fabry disease.
* Preferably two, but at minimum 1, historical serum creatinine evaluations in the last 2 years with the latest value within the last 6 months.
* Female patients and male patients whose co-partners are of child-bearing potential agree to use a medically acceptable method of contraception, not including the rhythm method. Acceptable methods of contraception include hormonal products, intrauterine device, or male or female condoms. Contraception should be used for 90 days after treatment discontinuation.

Exclusion Criteria:

* Patients enrolled and currently treated in Study PB-102-F20, and patients enrolled and currently treated in Extension Study PB-102-F60
* Patients who currently are on treatment under any other ongoing clinical trials of PRX-102
* History of Type 1 (anaphylaxis or anaphylactoid like) life-threatening hypersensitivity during previous exposure to other ERTs which could not be handled with medication
* Women who are breastfeeding may not participate unless they agree to stop breastfeeding.
* Women who are currently pregnant.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Inc., Phoenix, Arizona
  - University of California Irvine, Orange, California
  - Central Coas Nephrology, Salinas, California
  - University of Florida, Division of Pediatric Genetics, Jacksonville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Infusion Associates, Grand Rapids, Michigan
  - Dallas Nephrology Associates, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Lysosomal & Rare Disorder Research & Treatment Center (LRDRTC), Fairfax, Virginia